CLINICAL TRIAL: NCT01319513
Title: The Effect of the Pattern Post-exercise Aminoacidemia on Myofibrillar Protein Synthesis
Brief Title: Post-exercise Dietary Protein Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: RMIT University (Other); Australian Institute of Sport (Other); Nestec Ltd. (Industry)
Responsible Party: Dr. Stuart Phillips / Professor & Assoc. Chair Graduate Studies, McMaster University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Darwin 1a - Bolus versus Pulse
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Optimal Anabolic Nutrition Interventions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- protein feeding (Experimental): Participants will complete 2 trials in a cross-over fashion in which they will consume whey protein either as a single bolus or as 10 small divided doses
  Interventions: Other: whey protein bolus; Other: whey protein pulses

INTERVENTIONS:
Other: whey protein bolus — single dose of 25 g whey protein
Other: whey protein pulses — 10 2.5 g pulses of whey protein

SUMMARY:
Protein ingestion increases the rate at which the body builds new proteins in skeletal muscle (muscle protein synthesis. This study is designed to examine how the pattern of feeding affects muscle protein synthesis following resistance exercise. There is reason to believe that the large rapid increase in blood amino acid concentrations that accompanies the ingestion of a bolus of protein is important to increasing muscle protein synthesis. Thus, we hypothesize that the consumption a bolus of protein will elevate muscle protein synthesis to a greater extent than the consumption of an equivalent amount of protein that is consumed in small divided doses.

DETAILED DESCRIPTION:
The rapid appearance into the blood of essential amino acids, and leucine in particular, may act as an important signal to stimulate muscle protein synthesis after resistance exercise. This may explain why consuming rapidly-absorbed whey protein may have an anabolic edge over slowly-absorbed proteins such as casein. Previous investigations into importance of the rate of absorption to muscle protein synthesis that have used 'fast' and 'slow' proteins have been confounded by differences in amino acid composition. The present study addresses this issue by administering the same protein source, whey, as either a bolus or in small divided 'pulse' doses to achieve divergent amino acid profiles after a bout of resistance exercise.

This study is being conducted in young (18-35) men.

Our outcome measures include: blood amino acid concentrations, rates of myofibrillar protein synthesis, anabolic intracellular signalling markers

ELIGIBILITY:
Inclusion Criteria:

* Non-obese men (BMI <27) between the age of 18 and 35 yrs.

Exclusion Criteria:

* Type II diabetes or other known diseases
* Use of medication
* Female
* Other ages or BMI than indicated above
* Resistance training > 3X/wk

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Rate of myofibrillar protein synthesis | 4 months
  Rates of myofibrillar protein synthesis will be measured from muscle biopsy samples obtained from subjects participating in the study protocol.

SECONDARY OUTCOMES:
Myocellular protein phosphorylation | 4 months
  Protein phosphorylation of target proteins will be measured from Western blot analysis of muscle biopsy samples.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- Ivor Wynne Centre A103, McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] West DW, Burd NA, Coffey VG, Baker SK, Burke LM, Hawley JA, Moore DR, Stellingwerff T, Phillips SM. Rapid aminoacidemia enhances myofibrillar protein synthesis and anabolic intramuscular signaling responses after resistance exercise. Am J Clin Nutr. 2011 Sep;94(3):795-803. doi: 10.3945/ajcn.111.013722. Epub 2011 Jul 27. PMID 21795443